CLINICAL TRIAL: NCT01910415
Title: A Phase 1, Randomized, Placebo and Active Controlled, Double-Blind, Parallel, Electrocardiogram Study to Evaluate the Effect of Lumacaftor in Combination With Ivacaftor on the QT/QTc Interval in Healthy Subjects
Brief Title: Phase 1, QT/QTC Interval Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: VX12-809-008
Record Dates: First submitted 2013-07-19; First posted 2013-07-29 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Will consist of up to 4 cohorts with subjects receiving lumacaftor or placebo for 7 days.
  Cohort 1: 600 mg lumacaftor once a day Cohort 2: 1000 mg lumacaftor once a day Cohort 3: 1200 mg lumacaftor once a day
  Interventions: Drug: Lumacaftor; Drug: Lumacaftor Placebo
- Part B (Experimental): Will consist of 3 cohorts. All cohorts will be dosed in parallel. Cohort A will receive 600 mg Lumacaftor once a day plus 250 mg Ivacaftor twice a day for 7 days. From day 8-14 subjects will receive a supratherapeutic dose of Lumacaftor (TBD) plus 450 mg Ivacaftor twice a day.
  Cohort B will receive lumacaftor and ivacaftor matching placebo for 14 days Cohort C will receive a single dose of 400 mg moxifloxacin on day 14
  Interventions: Drug: Lumacaftor; Drug: Lumacaftor Placebo; Drug: Ivacaftor; Drug: Ivacaftor Placebo; Drug: moxifloxacin hydrochloride

INTERVENTIONS:
Drug: Lumacaftor
  Other Names: VX-809
Drug: Lumacaftor Placebo
Drug: Ivacaftor
  Other Names: VX-770
  Arms: Part B
Drug: Ivacaftor Placebo
  Arms: Part B
Drug: moxifloxacin hydrochloride
  Arms: Part B

SUMMARY:
This study is designed to evaluate the effect of multiple doses of lumacaftor in combination with ivacaftor on cardiac repolarization, as detected by QT/QTc interval corrected for heart rate in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to comply with scheduled visits, treatment plan, lifestyle guidelines, laboratory tests, contraceptive guidelines, and other study procedures.
* Subjects must be healthy, as defined by no clinically relevant abnormalities identified by a detailed medical history, physical examination, including blood pressure and pulse rate measurement, and 12 lead ECG.
* Subjects must weigh >50kg

Exclusion Criteria:

* Abnormal renal function at Screening
* Plasma donation within 7 days before first study drug dose or blood donation of 1 pint (500mL) within 56 days before first study drug dose
* Positively screen for Hepatitis B, Hepatitis C, HIV
* Known hypersensitivity or prior adverse reaction to moxifloxacin or other quinolones
* Any condition possibly affecting drug absorption (e.g., gastrectomy, or other gastrointestinal tract surgery, except appendectomy or cholecystectomy or polypectomy) or regular use of acid-lowering therapies (H2 blockers, proton pump inhibitors, and antacids).
* Female subjects who are pregnant, nursing, or planning to become pregnant during the study or within 90 days of the last study drug dose and female subjects of childbearing potential who are unwilling or unable to follow the contraceptive guidelines from at least 14 days before the first study drug dose.
* Male subject who has a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days of the last study drug dose; male subjects who are unwilling or unable to follow the contraceptive guidelines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
(Part A) Safety and tolerability of lumacaftor as measured by standard 12-lead ECGs, adverse events (AEs), vital signs, spirometry, and clinically significant laboratory assessments | 7 days
(Part B) Time matched, baseline-adjusted change in QTcF intervals obtained from a continuous ECG recording over a 24 hour interval after administration of a therapeutic and supratherapeutic dose of lumacaftor in combination with ivacaftor | 7 days

SECONDARY OUTCOMES:
(Part A) PK parameters of lumacaftor and M28-lumacaftor in plasma including Cmax and AUC | up to 11 days
(Part B) Time-matched, baseline-adjusted QTcF intervals obtained after a single 400-mg dose of moxifloxacin | up to 14 days
(Part B) Time-matched, baseline-adjusted non-QT interval parameters obtained from a continuous ECG recording over a 24-hour interval | up to 14 days
(Part B) PK parameters of lumacaftor, M28-lumacaftor, ivacaftor, M1-ivacaftor, and M6-ivacaftor including Cmax and AUC | up to 15 days
(Part B) PK/PD relationship between plasma concentration and QT/QTc interval | up to 14 days
(Part B) Safety and tolerability of lumacaftor in combination with ivacaftor as measured by standard 12-lead ECGs, AEs, vital signs, and clinical significant laboratory results | up to 24 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zuidlaren, Netherlands